CLINICAL TRIAL: NCT07341178
Title: Clinical Trial on Rapid Effects on Stem Cell Surveillance. A Randomized Placebo-controlled Acute Cross-over Trial.
Brief Title: Acute Effects on Stem Cell Surveillance
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Immune Systems Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 211-002
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Stem Cell Surveillance
Keywords: Stem cells; Flow cytometry; Surveillance; Mobilization; Homing
MeSH Terms: interventions — Fruit

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled, acute cross-over study design.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Crossover Group 1, randomized (Experimental): Participants consume a test product on each of the four clinic days, at least 1 week apart, allowing for 1 week wash-out period between each product. Participants will consume each of the 3 active test products versus placebo over 5 weeks, in this order: A, B, C, D.
  Interventions: Dietary Supplement: Anthocyanin-rich berry extract; Dietary Supplement: Anthocyanin-rich flower/leaf extract; Dietary Supplement: Berry /leaf blend; Dietary Supplement: Placebo
- Crossover Group 2, randomized (Experimental): Participants consume a test product on each of the four clinic days, at least 1 week apart, allowing for 1 week wash-out period between each product. Participants will consume each of the 3 active test products versus placebo over 5 weeks, in this order: B, C, D, A.
  Interventions: Dietary Supplement: Anthocyanin-rich berry extract; Dietary Supplement: Anthocyanin-rich flower/leaf extract; Dietary Supplement: Berry /leaf blend; Dietary Supplement: Placebo
- Crossover Group 3, randomized (Experimental): Participants consume a test product on each of the four clinic days, at least 1 week apart, allowing for 1 week wash-out period between each product. Participants will consume each of the 3 active test products versus placebo over 5 weeks, in this order: C, D. A, B.
  Interventions: Dietary Supplement: Anthocyanin-rich berry extract; Dietary Supplement: Anthocyanin-rich flower/leaf extract; Dietary Supplement: Berry /leaf blend; Dietary Supplement: Placebo
- Crossover Group 4, randomized (Experimental): Participants consume a test product on each of the four clinic days, at least 1 week apart, allowing for 1 week wash-out period between each product. Participants will consume each of the 3 active test products versus placebo over 5 weeks, in this order: D, A, B, C.
  Interventions: Dietary Supplement: Anthocyanin-rich berry extract; Dietary Supplement: Anthocyanin-rich flower/leaf extract; Dietary Supplement: Berry /leaf blend; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Anthocyanin-rich berry extract — 0.5 grams
Dietary Supplement: Anthocyanin-rich flower/leaf extract — 0.5 grams
Dietary Supplement: Berry /leaf blend — 0.5 grams
Dietary Supplement: Placebo — Placebo (white rice-based)

SUMMARY:
The goal for this clinical trial is to compare acute immune effects of three nutraceutical ingredients and blends to a placebo.

DETAILED DESCRIPTION:
The goal for this clinical trial is to compare acute immune effects of anthocyanin-rich botanical extracts and blends to a placebo.

Stem cell mobilization and homing will be evaluated through monitoring of changes to the numbers of various types of stem cells in the blood circulation.

The testing will show whether consuming the active test products lead to changes in stem cell numbers in circulation above the normal circadian changes for each participant. The normal circadian changes are documented on the clinic visit where placebo is consumed. Several different stem cell populations will be evaluated using flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults;
* Age 18-75 years (inclusive);
* Veins easy to see in one or both arms (to allow for the multiple blood draws);
* Willing to comply with study procedures, including:

  * Maintaining a consistent diet and lifestyle routine throughout the study,
  * Consistent habit of bland breakfasts on days of clinic visits,
  * Abstaining from exercising and nutritional supplements on the morning of a study visit,
  * Abstaining from use of coffee, tea, and soft drinks for at least one hour prior to a clinic visit,
  * Abstaining from music, candy, gum, computer/cell phone use, during clinic visits.

Exclusion Criteria:

* Previous major gastrointestinal surgery (absorption of test product may be altered) (minor surgery not a problem, including previous removal of appendix and gall bladder);
* Taking anti-inflammatory medications on a daily basis;
* Currently experiencing intense stressful events/ life changes;
* Currently in intensive athletic training (such as marathon runners);
* Currently taking anxiolytic, hypnotic, or anti-depressant prescription medication;
* An unusual sleep routine (examples: working graveyard shift, irregular routine with frequent late nights, studying, partying);
* Unwilling to maintain a constant intake of supplements over the duration of the study;
* Anxiety about having blood drawn;
* Pregnant, nursing, or trying to become pregnant;
* Known food allergies related to ingredients in active test product or placebo.

Prescription medication will be evaluated on a case-by-case basis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Stem cell surveillance | Baseline, 1 hour, 2 hours after consumption
  Changes to the number of stem cells in the blood circulation (number of cells per mL blood).
  Data is collected on the following types of stem cells: CD45dimCD34+CD309+, CD45dimCD34+CD309-, CD31++CD34-, CD45-CD90+.

SECONDARY OUTCOMES:
Serum cytokine levels | Baseline, 1 hour, 2 hours after consumption

CONTACTS AND LOCATIONS:
Locations (1):
- NIS Labs, Klamath Falls, Oregon, United States

IPD SHARING:
Plan to Share IPD: No